CLINICAL TRIAL: NCT06767410
Title: A Multi-domain Intervention to Constrast Cognitive Decline in Healthy Aging
Brief Title: A Multi-domain Intervention for Healthy Aging
Acronym: MultiMusic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Elvira Brattico, Professor, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ET-23-27
Record Dates: First submitted 2024-12-23; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteer Study
Keywords: BDNF; aging; multidomain intervention; music training; neuroplasticity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Multidomain group (Experimental): Participants who undergo regularly a series of activities involving different domains (e.g., physical activity, choir, horticulture etc.).
  Interventions: Other: Multidomain Intervention
- Active control group (Active Comparator): Participants who undergo regularly a series of activities but not musical acivities
  Interventions: Other: General activities
- Passive control group (No Intervention): Participants who undergo any activity or just sporadic activities

INTERVENTIONS:
Other: Multidomain Intervention — The intervention is distinguished by its multidomain approach combining cognitive, social, and musical activities through choir participation, targeting holistic cognitive and emotional benefits, unlike active controls (general activities) and passive controls (no activities).
  Arms: Multidomain group
Other: General activities — Participants will carry out a series of physical, manual and/or intellectual activities (e.g., horticulture, physical activities, theatre, learning programs etc.) but not musical activities
  Arms: Active control group

SUMMARY:
This study aims to investigate the long-term impact of a non-pharmacological intervention including several activities (e.g., physical activity, choir, learning programs, horticulture, etc.) to prevent cognitive impairment in community-dwelling elderly individuals with aspects of frailty. The main questions it aims to answer are:

* Does engaging in multiple activities, including music, slow the degeneration of perceptual and cognitive functions?
* Is it possible to foster beneficial brain changes even during aging?
* Can regularly attending social contexts reduce the risk of loneliness and provide fulfillment in later life? Researchers will compare participants involved in the multidomain intervention, including music, to another active group carrying out several activities but without music, and to a passive control group.

Participants will:

* Participate in the programs for 9 months;
* Be tested three times (before and after the intervention, and at a 6-month follow-up);
* Keep a weekly diary of the actual time spent in their activities.

DETAILED DESCRIPTION:
Brain-Derived Neurotrophic Factor (BDNF) plays a crucial role in neuroplasticity, supporting brain health throughout life and even during aging. This longitudinal study investigates the impact of a 9-month multidomain intervention, including choral practice, on BDNF levels, as well as audiometric and neuropsychological outcomes, in older adults, who are also assessed for their multidimensional frailty, based on their physical, cognitive, and nutritional conditions. BDNF levels, along with geriatric, neuropsychological, audiometric, and neurophysiological measures, are collected via saliva samples both pre- and post-intervention. For the longitudinal analyses of BDNF, up to 60 elderly individuals will be recruited from several recreational centers located in Southern Italy. Of these, one group will engage in a multidomain program that includes choir, physical, intellectual, and manual activities. The other two control groups will engage either in sporadic non-musical activities or no activity, or in various non-musical activities. Participation in all activities will be monitored via diaries.

The researchers' primary goal is to investigate whether engaging in physical, cognitive, and social activities can enhance neuroplasticity, as measured by BDNF levels, to counteract aspects of multidimensional frailty (as assessed by the multidimensional prognostic score, MPI) in the aging population. Secondly, the researchers aim to relate changes in BDNF levels to perceptual and cognitive functions and psychosocial well-being. Although previous studies point out the positive effects of musical training and active aging on brain health, the scarcity of longitudinal research on BDNF effects in older individuals leaves the issue open. Moreover, the researchers aim to test whether non-invasive, accessible saliva-based BDNF measurements, despite some reliability limitations, could offer indications of neuroprotection in aging.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65
* Living independently

Exclusion Criteria:

* Musical expertise
* Severe cognitive or functional impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Brain-Derived Neurotrophic Factor (BDNF) | Baseline, 9 months and 6 months follow-up
  BDNF levels detected in saliva
Cognitive functioning | Baseline, 9 months and 6 months follow-up
  Assessed using the Montreal Cognitive Assessment (MoCA) (Nasreddine et al., 2005), a widely used screening tool for cognitive impairment that evaluates multiple cognitive domains, including attention, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
  Description of the task:
  The MoCA consists of 30 items, covering various cognitive tasks such as word recall, trail-making, and visuospatial exercises.
  Unit of Measure:
  Raw score, ranging from 0 to 30, where higher scores indicate better cognitive functioning. A score below 26 typically indicates mild cognitive impairment.
  Interpretation:
  Higher scores reflect better cognitive performance. The measure is commonly used to detect cognitive deficits and track cognitive changes over time.
Fluid Intelligence | Baseline, 9 months and 6 months follow-up
  Assessed with computerized Matrix Reasoning (Condon & Revelle 2014; Chan & Kosinski, 2015), a test that contains stimuli that are similar to those used in Raven's Progressive Matrices.
  Task Description:
  The stimuli are 3 × 3 arrays of geometric shapes with one of the nine shapes missing. Participants are instructed to identify which of the six geometric shapes presented as response choices will best complete the stimuli. In each round the stimulus disappears after 120 s, leaving only the response options visible for the participant.
  Unit of Measure:
  The score is calculated as a standardized z-score, with a mean of 0 and no fixed minimum or maximum value. Scores can be both positive or negative, depending on the participant's performance relative to the sample distribution.
  Interpretation:
  Higher positive scores indicate better-than-average performance in reasoning ability, while negative scores indicate below-average performance. This measure is suitable for evaluating individual
Hearing Threshold | Baseline, 9 months and 6 months follow-up
  Assessed using a liminal tonal audiometric test, which determines the participant's minimum acoustic intensity perceivable at different tonal field frequencies.
  Description of the task:
  Participants are tested across a range of frequencies in a soundproof booth to identify the lowest intensity level at which they can detect a tone.
  Unit of Measure:
  Hearing threshold in decibels hearing level (dB HL), measured for each frequency. Lower thresholds (i.e., lower dB HL values) indicate better hearing sensitivity.
  Interpretation:
  Lower dB HL values indicate better hearing ability. The results are used to identify any hearing loss and its severity at specific frequencies.
Intelligibility | Baseline, 9 months and 6 months follow-up
  Assessed using speech audiometry, which evaluates the participant's ability to recognize and understand spoken words in a controlled environment.
  Description of the task:
  Participants are presented with vocal material (e.g., phonemes, logotomes, words, sentences) in a silent booth and must repeat what they hear.
  Unit of Measure:
  Percentage of correctly recognized words, where higher percentages indicate better speech intelligibility.
  Interpretation:
  Higher percentages indicate better verbal recognition and understanding. This measure helps assess speech comprehension in quiet conditions.
Speech in noise ability | Baseline, 9 months and 6 months follow-up
  Assessed using a Matrix Sentence Test, which evaluates speech comprehension under noisy conditions.
  Description of the task:
  Participants are presented with 5-word sentences along with a background noise (competition noise) and must repeat the sentences. The test adapts after each response by adjusting the difficulty (increasing or decreasing the noise level) until the participant reaches a 50% comprehension threshold.
  Unit of Measure:
  Signal Reception Threshold (SRT) in decibels (dB). The SRT represents the difference between the word volume and the noise volume at which the participant understands 50% of the words.
  Interpretation:
  Lower SRT values indicate better speech comprehension under noisy conditions.
Auditory brainstem responses (ABR) | Baseline, 9 months and 6 months follow-up
  Measure of the neural activity along the auditory pathway in response to a brief acoustic stimulus.
  Description of the task:
  Short-duration acoustic stimuli (100 μs clicks) are presented independently to each ear at 90 dBnHL, with filters set at 100 and 3000 Hz. The resulting waveforms represent the activity of the auditory nerve and brainstem.
  Unit of Measure:
  Latencies of waves I-V in milliseconds (ms). Longer latencies may indicate abnormalities in the auditory pathway.
  Interpretation:
  Normal latencies indicate typical auditory nerve and brainstem function. Abnormal latencies may suggest issues such as hearing loss or neural conduction delays.
P300 auditory cortical potentials | Baseline, 9 months and 6 months follow-up
  Measures higher-level auditory processing and cognitive responses to auditory stimuli.
  Description of the task:
  Tones (50 ms) are presented at a rate of 1.1/s, with standard stimuli occurring 80% of the time and target stimuli randomly occurring 20% of the time. Participants are required to detect and respond to the target stimuli. The P300 response is recorded using electrodes in the same montage as for the ABR.
  Unit of Measure:
  P300 latency in milliseconds (ms) and P300 amplitude in microvolts (µV). Shorter latencies and higher amplitudes indicate better cognitive and auditory processing.
  Interpretation:
  Shorter P300 latencies and higher amplitudes suggest more efficient auditory and cognitive processing. Prolonged latencies or reduced amplitudes may indicate deficits in auditory or cognitive functions.
Multidimensional Frailty | Baseline, 9 months and 6 months follow-up
  Assessed using the Selfy-MPI (Pilotto et al., 2019), a self-administered digital tool via the Portable-MPI app.
  Description:
  The Selfy-MPI evaluates frailty across several dimensions, including:
  Functional status and independence: Measured by ADLs and IADLs.
  Mobility: Assessed through self-reported ability to move independently.
  Cognitive condition: Evaluated with a brief cognitive test.
  Nutritional status: Measured using the Mini Nutritional Assessment (MNA).
  Comorbidity: Assessed using the Cumulative Illness Rating Scale (CIRS).
  Medication use: Evaluated via the ATC classification for polypharmacy.
  Living situation: Assessed by questions on living arrangements.
  Unit of Measure:
  Composite score ranging from 0 to 1, where:
  0-0.33: Low frailty risk 0.34-0.66: Moderate frailty risk 0.67-1.00: Severe frailty risk
  Interpretation:
  Higher scores indicate greater frailty.
Socio-psychological well being | Baseline, 9 months and 6 months follow-up
  Assessed using the Flourishing Scale (Diener et al., 2010), a self-report measure that evaluates various domains, including relationships, purpose in life, and self-esteem.
  Description of the task:
  Participants rate 8 statements related to different aspects of their well-being (e.g., "I lead a purposeful and meaningful life") on a scale from 1 (Strongly disagree) to 7 (Strongly agree).
  Unit of Measure:
  The total score ranges from 8 to 56, with higher scores indicating greater psychological flourishing and well-being.
  Interpretation:
  Higher scores reflect better overall well-being, life satisfaction, and psychological functioning.

SECONDARY OUTCOMES:
Physical activity | Baseline, 9 months and 6 months follow-up
  Assessed using the Global Physical Activity Questionnaire (GPAQ), developed by Armstrong & Bull (2006) for the World Health Organization (WHO) to measure physical activity levels across different domains of daily life.
  Description of the task:
  The GPAQ collects self-reported information on physical activity in three domains:
  Work-related physical activity Travel to and from places (active transport) Recreational physical activity It also includes a section on sedentary behavior.
  Unit of Measure:
  Physical activity is reported in Metabolic Equivalent of Task (MET) minutes per week.
  Sedentary behavior is reported in minutes per day spent sitting.
  Interpretation:
  Higher MET minutes indicate greater physical activity levels, while higher sedentary minutes indicate lower activity and greater sedentary behavior.
Cognitive Reserve | Baseline, 9 months and 6 months follow-up
  Assessed using the Cognitive Reserve Index Questionnaire (CRIq), developed by Nucci, Mapelli & Mondini (2012), a tool designed to estimate an individual's cognitive reserve based on their lifetime activities.
  Description of the task:
  The CRIq collects self-reported information across three domains:
  Education (CRI-E): Years of formal education and training. Working activity (CRI-W): Type and duration of work experience, categorized by cognitive demand.
  Leisure time activities (CRI-L): Participation in cognitively stimulating activities during leisure time (e.g., reading, social engagement, cultural activities).
  Unit of Measure:
  The questionnaire provides a total Cognitive Reserve Index (CRI) score, along with sub-scores for each domain (CRI-E, CRI-W, CRI-L). The total score is standardized, with higher values indicating greater cognitive reserve.
  Interpretation:
  Higher CRI scores suggest a higher level of cognitive reserve, which is associated with better cognitive functioning and r
Melody Discrimination | Baseline, 9 months and 6 months follow-up
  Assessed using the Melody Discrimination Test (MDT), an adaptive task based on a three-alternative forced-choice (3-AFC) melodic discrimination paradigm, developed by Harrison et al. (2017). The test evaluates participants' ability to discriminate between similar melodies by identifying the melody with a single altered note.
  Description of the task:
  In each trial, participants hear three versions of the same melody. Two of the versions (lures) have the same interval structure, while the third version (the odd-one-out) contains a single altered note.
  Participants are required to identify the odd-one-out melody by first identifying the most similar pair and then selecting the melody that is different.
  The difficulty of the items is adaptively adjusted by manipulating the length of the melodies. In this study, the test consists of 18 items.
  Unit of Measure:
  Standardized z-score, with a mean of 0 and no fixed minimum or maximum value. Scores can be positive or negative, depending on the
Mistuning Perception | Baseline, 9 months and 6 months follow-up
  Assessed using the Mistuning Perception Test (MPT) (Larrouy-Maestri et al., 2019), which evaluates the ability to detect mistuning in musical extracts.
  Description of the task: In each trial, participants are presented with two versions of a musical excerpt-one "in tune" and one "out of tune"-and must identify the out-of-tune version. The stimulus material consists of short excerpts (6-12 s in length) from pop music performances (obtained from MedleyDB; Bittner et al., 2017) for which the vocal track was pitch-shifted relative to the instrumental tracks. Each musical extract has a vocalist singing the main melodic line and an instrumental accompaniment. Out-of-tune extracts are produced by adding a constant pitch shift to the vocal line
  Unit of Measure:
  Standardized z-score with a mean of 0, where scores can be positive or negative.
  Interpretation:
  Higher scores indicate better mistuning perception.
Emotion Discrimination | Baseline, 9 months and 6 months follow-up
  Assessed using the Emotion Discrimination Test (EDT) (MacGregor & Müllensiefen, 2019), an adaptive test that evaluates the ability to distinguish emotions conveyed by musical fragments.
  In each trial, participants are presented with two versions of a melody and must identify which fragment corresponds to a specific target emotion (anger, happiness, sadness, or tenderness). Excerpts differ between trials in terms of musical features such as length, instrument, melody, target emotion and comparison emotion, and item difficulty is assessed with regard to the contribution of these features.
  Unit of Measure:
  Standardized z-score, with a mean of 0, where scores can be positive or negative.
  Interpretation:
  Higher scores indicate better ability to discriminate emotions in music.
Rhythmic Ability | Baseline, 9 months and 6 months follow-up
  Assessed using the Rhythm Ability Test (RAT) (MacGregor et al., 2022), an adaptive test that evaluates rhythmic perception. Participants hear a rhythm composed of high-pitched and low-pitched sounds and must select the image that correctly represents the rhythm, where sounds are visually indicated by squares of different colors in two rows.
  Description of the task:
  The rhythms are made up of high-pitched and low-pitched sounds. High-pitched and low-pitched sounds are represented in each picture with two rows of squares of two different colors placed at the top row (to indicate high-pitched sounds) and at the bottom row (to indicate low-pitched sounds). The tasks are presented according to a progressive increasing difficulty, and the stimuli are made up of 4, 8, and 16 sounds (quarter, eights, sixteenths notes).
  Unit of Measure:
  Standardized z-score, with a mean of 0, where scores can be positive or negative.
  Interpretation:
  Higher scores indicate better rhythmic ability.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Musica In Gioco, Adelfia, Bari
  - University of Bari, Bari, Bari
  - Centro Servizi per la famiglia Libertà, Bari, Bari
  - ANAS Puglia (Associazione Nazionale di Azione Sociale), Bari, Bari

IPD SHARING:
Plan to Share IPD: Yes
We will share anonymized derived data, including salivary BDNF levels and neurophysiological data, but not the biological saliva samples due to logistical limitations, ethical constraints regarding participant consent, and the adequacy of the derived data to support further analyses. This ensures transparency while respecting ethical and practical considerations.

REFERENCES:
- [Background] Wang X, Soshi T, Yamashita M, Kakihara M, Tsutsumi T, Iwasaki S, Sekiyama K. Effects of a 10-week musical instrument training on cognitive function in healthy older adults: implications for desirable tests and period of training. Front Aging Neurosci. 2023 Aug 15;15:1180259. doi: 10.3389/fnagi.2023.1180259. eCollection 2023. PMID 37649718
- [Background] Vrijen C, Schenk HM, Hartman CA, Oldehinkel AJ. Measuring BDNF in saliva using commercial ELISA: Results from a small pilot study. Psychiatry Res. 2017 Aug;254:340-346. doi: 10.1016/j.psychres.2017.04.034. Epub 2017 Apr 22. PMID 28525789
- [Background] Veronese N, Noale M, Cella A, Custodero C, Smith L, Barbagelata M, Maggi S, Barbagallo M, Sabba C, Ferrucci L, Pilotto A. Multidimensional frailty and quality of life: data from the English Longitudinal Study of Ageing. Qual Life Res. 2022 Oct;31(10):2985-2993. doi: 10.1007/s11136-022-03152-9. Epub 2022 May 17. PMID 35579730
- [Background] Seinfeld S, Figueroa H, Ortiz-Gil J, Sanchez-Vives MV. Effects of music learning and piano practice on cognitive function, mood and quality of life in older adults. Front Psychol. 2013 Nov 1;4:810. doi: 10.3389/fpsyg.2013.00810. eCollection 2013. PMID 24198804
- [Background] Rosenberg A, Ngandu T, Rusanen M, Antikainen R, Backman L, Havulinna S, Hanninen T, Laatikainen T, Lehtisalo J, Levalahti E, Lindstrom J, Paajanen T, Peltonen M, Soininen H, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Solomon A, Kivipelto M. Multidomain lifestyle intervention benefits a large elderly population at risk for cognitive decline and dementia regardless of baseline characteristics: The FINGER trial. Alzheimers Dement. 2018 Mar;14(3):263-270. doi: 10.1016/j.jalz.2017.09.006. Epub 2017 Oct 19. PMID 29055814
- [Background] Perus L, Busto GU, Mangin JF, Le Bars E, Gabelle A. Effects of preventive interventions on neuroimaging biomarkers in subjects at-risk to develop Alzheimer's disease: A systematic review. Front Aging Neurosci. 2022 Nov 24;14:1014559. doi: 10.3389/fnagi.2022.1014559. eCollection 2022. PMID 36506466
- [Background] Pentikainen E, Kimppa L, Pitkaniemi A, Lahti O, Sarkamo T. Longitudinal effects of choir singing on aging cognition and wellbeing: a two-year follow-up study. Front Hum Neurosci. 2023 Jul 20;17:1174574. doi: 10.3389/fnhum.2023.1174574. eCollection 2023. PMID 37545597
- [Background] Nazam F, Shaikh S, Nazam N, Alshahrani AS, Hasan GM, Hassan MI. Mechanistic insights into the pathogenesis of neurodegenerative diseases: towards the development of effective therapy. Mol Cell Biochem. 2021 Jul;476(7):2739-2752. doi: 10.1007/s11010-021-04120-6. Epub 2021 Mar 9. PMID 33687588
- [Background] Nettiksimmons J, Simonsick EM, Harris T, Satterfield S, Rosano C, Yaffe K; Health ABC Study. The associations between serum brain-derived neurotrophic factor, potential confounders, and cognitive decline: a longitudinal study. PLoS One. 2014 Mar 26;9(3):e91339. doi: 10.1371/journal.pone.0091339. eCollection 2014. PMID 24670553
- [Background] Moon SY, Kim S, Choi SH, Hong CH, Park YK, Na HR, Song HS, Park HK, Choi M, Lee SM, Chun BO, Lee JM, Jeong JH. Impact of Multidomain Lifestyle Intervention on Cerebral Cortical Thickness and Serum Brain-Derived Neurotrophic Factor: the SUPERBRAIN Exploratory Sub-study. Neurotherapeutics. 2022 Sep;19(5):1514-1525. doi: 10.1007/s13311-022-01276-x. Epub 2022 Aug 1. PMID 35915368
- [Background] Mizoguchi Y, Yao H, Imamura Y, Hashimoto M, Monji A. Lower brain-derived neurotrophic factor levels are associated with age-related memory impairment in community-dwelling older adults: the Sefuri study. Sci Rep. 2020 Oct 5;10(1):16442. doi: 10.1038/s41598-020-73576-1. PMID 33020545
- [Background] Marie D, Muller CAH, Altenmuller E, Van De Ville D, Junemann K, Scholz DS, Kruger THC, Worschech F, Kliegel M, Sinke C, James CE. Music interventions in 132 healthy older adults enhance cerebellar grey matter and auditory working memory, despite general brain atrophy. Neuroimage Rep. 2023 Mar 23;3(2):100166. doi: 10.1016/j.ynirp.2023.100166. eCollection 2023 Jun. PMID 40568451
- [Background] MacAulay, R. K., Edelman, P., Boeve, A., Sprangers, N., & Halpin, A. (2019). Group music training as a multimodal cognitive intervention for older adults. Psychomusicology: Music, Mind, and Brain, 29(4), 180.
- [Background] Lin FR, Ferrucci L, Metter EJ, An Y, Zonderman AB, Resnick SM. Hearing loss and cognition in the Baltimore Longitudinal Study of Aging. Neuropsychology. 2011 Nov;25(6):763-70. doi: 10.1037/a0024238. PMID 21728425
- [Background] Lee S, Harada K, Bae S, Harada K, Makino K, Anan Y, Suzuki T, Shimada H. A non-pharmacological multidomain intervention of dual-task exercise and social activity affects the cognitive function in community-dwelling older adults with mild to moderate cognitive decline: A randomized controlled trial. Front Aging Neurosci. 2023 Mar 13;15:1005410. doi: 10.3389/fnagi.2023.1005410. eCollection 2023. PMID 36993908
- [Background] Johnson JK, Louhivuori J, Stewart AL, Tolvanen A, Ross L, Era P. Quality of life (QOL) of older adult community choral singers in Finland. Int Psychogeriatr. 2013 Jul;25(7):1055-64. doi: 10.1017/S1041610213000422. Epub 2013 Apr 11. PMID 23574947
- [Background] Jabusch HC, Alpers H, Kopiez R, Vauth H, Altenmuller E. The influence of practice on the development of motor skills in pianists: a longitudinal study in a selected motor task. Hum Mov Sci. 2009 Feb;28(1):74-84. doi: 10.1016/j.humov.2008.08.001. Epub 2008 Oct 8. PMID 18845349
- [Background] Huang TY, Chou MY, Liang CK, Lin YT, Chen RY, Wu PF. Physical activity plays a crucial role in multidomain intervention for frailty prevention. Aging Clin Exp Res. 2023 Jun;35(6):1283-1292. doi: 10.1007/s40520-023-02412-z. Epub 2023 Apr 26. PMID 37101084
- [Background] Hariri AR, Goldberg TE, Mattay VS, Kolachana BS, Callicott JH, Egan MF, Weinberger DR. Brain-derived neurotrophic factor val66met polymorphism affects human memory-related hippocampal activity and predicts memory performance. J Neurosci. 2003 Jul 30;23(17):6690-4. doi: 10.1523/JNEUROSCI.23-17-06690.2003. PMID 12890761
- [Background] Ellis RJ, Bruijn B, Norton AC, Winner E, Schlaug G. Training-mediated leftward asymmetries during music processing: a cross-sectional and longitudinal fMRI analysis. Neuroimage. 2013 Jul 15;75:97-107. doi: 10.1016/j.neuroimage.2013.02.045. Epub 2013 Mar 5. PMID 23470982
- [Background] Egan MF, Kojima M, Callicott JH, Goldberg TE, Kolachana BS, Bertolino A, Zaitsev E, Gold B, Goldman D, Dean M, Lu B, Weinberger DR. The BDNF val66met polymorphism affects activity-dependent secretion of BDNF and human memory and hippocampal function. Cell. 2003 Jan 24;112(2):257-69. doi: 10.1016/s0092-8674(03)00035-7. PMID 12553913
- [Background] Dubinsky E, Wood EA, Nespoli G, Russo FA. Short-Term Choir Singing Supports Speech-in-Noise Perception and Neural Pitch Strength in Older Adults With Age-Related Hearing Loss. Front Neurosci. 2019 Nov 28;13:1153. doi: 10.3389/fnins.2019.01153. eCollection 2019. PMID 31849572
- [Background] Driscoll I, Martin B, An Y, Maudsley S, Ferrucci L, Mattson MP, Resnick SM. Plasma BDNF is associated with age-related white matter atrophy but not with cognitive function in older, non-demented adults. PLoS One. 2012;7(4):e35217. doi: 10.1371/journal.pone.0035217. Epub 2012 Apr 16. PMID 22523577
- [Background] Draganski B, Gaser C, Busch V, Schuierer G, Bogdahn U, May A. Neuroplasticity: changes in grey matter induced by training. Nature. 2004 Jan 22;427(6972):311-2. doi: 10.1038/427311a. No abstract available. PMID 14737157
- [Background] Dichter BK, Breshears JD, Leonard MK, Chang EF. The Control of Vocal Pitch in Human Laryngeal Motor Cortex. Cell. 2018 Jun 28;174(1):21-31.e9. doi: 10.1016/j.cell.2018.05.016. PMID 29958109
- [Background] Chikahisa S, Sei H, Morishima M, Sano A, Kitaoka K, Nakaya Y, Morita Y. Exposure to music in the perinatal period enhances learning performance and alters BDNF/TrkB signaling in mice as adults. Behav Brain Res. 2006 May 15;169(2):312-9. doi: 10.1016/j.bbr.2006.01.021. Epub 2006 Mar 10. PMID 16530277
- [Background] Chaddock-Heyman L, Loui P, Weng TB, Weisshappel R, McAuley E, Kramer AF. Musical Training and Brain Volume in Older Adults. Brain Sci. 2021 Jan 5;11(1):50. doi: 10.3390/brainsci11010050. PMID 33466337
- [Background] Bugos JA, Perlstein WM, McCrae CS, Brophy TS, Bedenbaugh PH. Individualized piano instruction enhances executive functioning and working memory in older adults. Aging Ment Health. 2007 Jul;11(4):464-71. doi: 10.1080/13607860601086504. PMID 17612811
- [Background] Bugos JA, Bidelman GM, Moreno S, Shen D, Lu J, Alain C. Music and Visual Art Training Increase Auditory-Evoked Theta Oscillations in Older Adults. Brain Sci. 2022 Sep 27;12(10):1300. doi: 10.3390/brainsci12101300. PMID 36291234
- [Background] Bonetti L, Bruzzone SEP, Paunio T, Kantojarvi K, Kliuchko M, Vuust P, Palva S, Brattico E. Moderate associations between BDNF Val66Met gene polymorphism, musical expertise, and mismatch negativity. Heliyon. 2023 Apr 18;9(5):e15600. doi: 10.1016/j.heliyon.2023.e15600. eCollection 2023 May. PMID 37153429
- [Background] Alain C, Moussard A, Singer J, Lee Y, Bidelman GM, Moreno S. Music and Visual Art Training Modulate Brain Activity in Older Adults. Front Neurosci. 2019 Mar 8;13:182. doi: 10.3389/fnins.2019.00182. eCollection 2019. PMID 30906245